CLINICAL TRIAL: NCT02189850
Title: Efficacy, Safety and Tolerability of a Bowel Cleansing Preparation (BLI800) in Pediatric Subjects Undergoing Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLI800-501
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Colonoscopy
Keywords: colonoscopy; pediatric

ARMS (2):
- BLI800 - Dose 1 (Experimental): BLI800 oral solution
  Interventions: Drug: BLI800 - Dose 1
- BLI800 - Dose 2 (Experimental): BLI800 oral solution
  Interventions: Drug: BLI800 - Dose 2

INTERVENTIONS:
Drug: BLI800 - Dose 1 — BLI800 oral solution
  Other Names: BLI800
  Arms: BLI800 - Dose 1
Drug: BLI800 - Dose 2 — BLI800 oral solution
  Other Names: BLI800
  Arms: BLI800 - Dose 2

SUMMARY:
The purpose o this study is to evaluate the safety, tolerance and efficacy of BLI800 as a bowel preparation prior to colonoscopy in pediatric patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female between the ages of 12 to 17
* Weight more than 40kg
* Undergoing colonoscopy for routinely accepted indications
* If female, and of child-bearing potential, subject must use an acceptable form of birth control or remain abstinent for the duration of the study.
* Negative pregnancy test at screening, if applicable
* In the Investigator's judgment, caregiver is mentally competent to provide informed consent for their child to participate in the study.

Exclusion Criteria:

* Subjects with known or suspected ileus, impaction, severe ulcerative colitis, acute peritonitis, gastrointestinal obstruction, gastric retention (gastroparesis), bowel perforation, toxic colitis or megacolon.
* Subjects who had previous significant gastrointestinal surgeries.
* Subjects with increased risk of bowel perforation, including connective tissue disorders, toxic dilation of the bowel or recent bowel surgery.
* Subjects with uncontrolled pre-existing electrolyte abnormalities, or those with clinically significant electrolyte abnormalities based on Visit 1 laboratory results
* Subjects with bleeding disorders and/or impaired platelet function, or neutropenia.
* Subjects with a prior history of renal, liver or cardiac insufficiency
* Subjects required to take any other oral medication within 3 hours of dosing until completion of both doses.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects with tendency for nausea and/or vomiting, or that have known swallowing disorders.
* Subjects for whom intake of substances is likely to affect gastrointestinal motility or urinary flow rate.
* Subjects undergoing colonoscopy for foreign body removal and/or decompression.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - Delta Research Partners, Bastrop, Louisiana
  - Gastrointestinal Associates, Jackson, Mississippi
  - University of Buffalo Pediatric Associates, Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- BLI800 - Dose 1: BLI800 oral solution
  BLI800 - Dose 1: BLI800 oral solution (6 oz)
- BLI800 - Dose 2: BLI800 oral solution
  BLI800 - Dose 2: BLI800 oral solution (4.5 oz)
Period: Overall Study
Arm/Group | BLI800 - Dose 1 | BLI800 - Dose 2
Started (Safety population - all subjects that took preparation.) | 16 | 13
Completed | 14 | 11
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population - all subjects that took preparation.
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI800 - Dose 1 | BLI800 - Dose 2 | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.2) | 15.8 (1.4) | 15.5 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 9 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 29
Puburtal Staging [Count of Participants; unit: Participants] — Pubertal Tanner Staging from I (prepubertal) to V (adult genitalia)
  Participants
    I | 0 | 0 | 0
    II | 0 | 1 | 1
    III | 1 | 0 | 1
    IV | 3 | 1 | 4
    V | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: % of Subjects With Successful Preparation Rated by Colonoscopist on a 4 Point Scale (1=Poor to 4 = Excellent)
Description: Successful Preparation, defined as a colonoscopy rated as Excellent or Good by the blinded endoscopist.
  Poor: Large amounts of fecal residue, additional bowel preparation required; Fair: Enough feces even after washing and suctioning to prevent clear visualization of the entire colonic mucosa; Good: Feces and fluid requiring washing and suctioning, but still achieves clear visualization of the entire colonic mucosa; Excellent: No more than small bits of feces/fluid which can be suctioned easily; achieves clear visualization of the entire colonic mucosa
Time Frame: 2 days
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800 - Dose 1 | BLI800 - Dose 2
Number analyzed (Participants) | 16 | 12
Participants | 13 | 10
Statistical Analysis 1: Comparison: BLI800 - Dose 1 vs BLI800 - Dose 2; Test type: Superiority; p = 0.923, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Arm/Group | BLI800 - Dose 1 | BLI800 - Dose 2
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 13/16 | 12/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI800 - Dose 1 (N=16) | BLI800 - Dose 2 (N=13)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 4 (4)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 6 (6)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bacterial test (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Urinary casts (Investigations) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable